CLINICAL TRIAL: NCT03305952
Title: Cognitively-Based Compassion Training (CBCT) for the Improvement of Health Related Quality of Life, Fear of Illness Recurrence, Compassion and Self-compassion in Breast Cancer Survivors Sample
Brief Title: Cognitively-Based Compassion Training for Breast Cancer Survivors
Acronym: CBCT-BC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rosa María Baños Rivera, Full professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CBCT-IVO
Record Dates: First submitted 2017-10-02; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Compassion; Treatment as Usual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compassion (Experimental): CBCT was facilitated in an eight weekly, 2-h sessions format through didactics, class discussion, and guided meditation practice. Topics covered in order were: Week 1: Developing attention stability and mental clarity. Week 2. Open awareness of sensations, feelings, and emotions. Week 3: Self-Compassion. Week 4: Practice in impartiality and cultivation of social connection. Week 5: Practice in appreciation, gratitude, social interconnection, and interdependence. Session 6: Practice in affection (endearment) for developing undifferentiated affection for others. Week 7: Development of the aspirational wish that all beings be happy and free from suffering and its causes. Week 8: Active compassion
  Interventions: Behavioral: CBCT
- Treatment as usual (Active Comparator): Treatment as usual (TAU) consisted of usual periodical visits to psycho oncologist based on hospital's regular calendar. Hospital's standard treatment was applied to participants. The standard treatment consists of counselling interventions, cognitive-behavioural interventions, family interventions, third generation interventions.
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: CBCT
  Arms: Compassion
Other: TAU
  Arms: Treatment as usual

SUMMARY:
There is a growing number of evidence of how mindfulness training enhances psychological and physical well-being and coping strategies in patients with oncological illnesses. However, there are very few studies analyzing the efficacy of Compassion-Based Interventions on breast cancer survivors.

The goal of this study is to analyze enrollment, participant satisfaction and adherence to program and differences in psychological well-being, health related quality of life, fear of illness recurrence, compassion and self-compassion variables after a Compassion-Based Intervention in a Spanish breast cancer survivor sample.

This study is a randomized clinical trial of a secularized intervention called Cognitively-Based Compassion Training (CBCT). Subjects (n = 58) were randomly assigned to CBCT (n = 28) or a treatment as usual control group (TAU) (n = 28). Participants in the CBCT intervention condition were asked to meet weekly for a two (2) hour long session during two months. Pre-post-intervention and six month follow-up measures took place to evaluate: psychological well-being (somatic, depressive, and anxious symptomatology), health related quality of life (physical, social, emotional, and functional); psychological stress, coping strategies and triggering cognitions linked to cancer recurrence fear, self-compassion, compassion and mindfulness and awareness in both intervention and wait list groups.

CBCT is a promising and potentially useful intervention to enhance physical and emotional well-being in breast cancer survivors. Nevertheless, future randomized trials are needed and a process of cultural adaptation required.

DETAILED DESCRIPTION:
About 1 in 8 U.S. women (around 12%) will develop invasive Breast Cancer (BC) over the course of his/her lifetime. In 2015 there were 231,840 new cases of Breast Cancer (BC) in the United States and it is this type of cancer with more new cases from all the rest. In 2017, an estimated 252,710 new cases of invasive BC are expected to be diagnosed in women in the U.S., along with 63,410 new cases of non-invasive (in situ) BC. In Spain, there are around 21,000 new cases of BC every year. Among the different types of cancer, this is the one that shows higher incidence, mortality, and prevalence to 5 years (29%, 15.5%, and 40.8%, respectively).

Common to all organic illnesses, BC has a number of associated physical, social and psychological impairments, like problems of adaptation, difficulties in communication, or depressive and anxious symptoms. Psychological and emotional stress in patients increases the experience of pain, reduces the overall performance and is a fundamental factor of suicidal ideation and suicide attempts.

In addition to having to deal with intrusive medical procedures and treatment (chemotherapy and/or radiotherapy) side effects, BC patients treatment requires a significant psychological adaptation. Furthermore, once treatment is finished, the fear of cancer recurrence occurs in around 70% of the patients, which is associated with long-term functional impairments. In addition, in nearly half of the survivors, intrusive thoughts about the disease and its treatment (unwanted thoughts, images and memories) occur years after successful treatment. In such patients, it has been observed that even when the rates of depression decreased, overall well-being does not improve. Fatigue and sleep problems are also clinically significant in 60% of these kinds of patients, which creates imbalances both functional and in quality of life.

Nowadays there are many psychological interventions that have been shown to be beneficial for patients with BC. The most used and with a bigger body of evidence are those interventions of cognitive-behavioral nature. There are three areas where cognitive-behavioral interventions have had a greater impact on breast cancer patients' care: (1) treatment for pain relief; (2) control of the aversive reactions of chemotherapy; and (3) improvement of emotional well-being.

In recent years, interest in Mindfulness-Based Interventions (MBI) research for breast cancer patients has increased, especially for those who have passed the initial malignancy and its treatment, but often have to deal with functional, behavioral and persistent emotional difficulties, such as depression, fatigue, fear of illness recurrence and cognitive impairments. A Systematic review has shown positive results as an effective coping strategy that diminishes anxiety, stress, fatigue, general mood, sleep disturbances, and enhances quality of life.

Like Mindfulness, compassion can be trained using specific techniques and protocols (Compassion-Based Intervention, CBI) designed specifically for this purpose. As a matter of fact, for some authors CBIs may provide useful tools and resources to treat and prevent various types of psychological difficulties (resources for interpersonal relationships, reduction of depressive symptomatology, reduction of social anxiety, marital conflict, anger management and dealing with the difficulties of being a caregiver).

In one study authors found how a CBI was associated with decreasing innate immune responses to a psychosocial stressor. One research showed how loving-kindness (an ability often trained in CBIs) practice was associated with less pain during that whole day and lower anger during the next. Another study observed study observed how a CBI could significantly reduce the feeling of loneliness and increase positive emotions. Some authors found an increase in positive emotions in everyday experiences after training in compassion, which, in turn, enhanced personal resources (purpose in life, social connection, and decrease in disease symptoms). Although there are numerous studies on compassion and self-compassion in different types of healthy populations and in clinical settings, there are hardly any data on the benefits of CBIs in cancer patients.

Cognitively-Based Compassion Training (CBCT) is a secular protocol to teach compassion. The foundational technique that CBCT uses to bring about a shift in perspective is to ground the individual in a non-judgmental attentiveness to the present moment, followed by cognitive exercises or analytical meditations. CBCT Program has shown to be effective in reducing hormone levels related to psychoimmunological stress systems, as well as regulation of inflammatory processes in adolescent population with early life adverse events. Recently, a study found that CBCT program was a potentially effective and beneficial intervention and highly satisfactory for the psychological well-being of breast cancer survivors. Nevertheless, effects of CBCT on health-related quality of life, general well-being, mindfulness facets, self-compassion and compassion traits have not yet been shown.

The goal of this study was to analyze the efficacy of CBCT Protocol in a Randomized Clinical Trial (RCT) on a sample of breast cancer survivors over physical and psychological well-being (somatic, depressive, anxious symptomatology); health-related quality of life (physical, social, emotional and functional quality of life); psychological dimensions linked to fear of cancer recurrence, levels of Mindfulness facets, Self-Compassion and Compassion.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 35 and 75 years,
* Being able to read and write using the Spanish language,
* History of treated Breast Cancer within the past 15 years,
* Free from oncological illness
* Not receiving any kind of chemotherapy and / or radiotherapy treatment during study.

Eligible participants were contacted by their personal psychooncologist either by a telephone call or at psychooncology appointment periodical visit to invite them to an explanatory meeting of the study.

Exclusion Criteria:

* Active severe mental disorders (schizophrenia, bipolar disorder, eating disorders, and major depression),
* Substance use disorders, cognitive impairment,
* Impaired medical condition.

Past and current psychiatric and medical history was determined by clinician assessment with the Mini International Neuropsychiatric Interview (MINI) (Lecrubier et al., 1997) Spanish version (Lobo et al., 1999).

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-01-11 (Actual); Primary Completion 2018-07-18 (Estimated); Study Completion 2018-07-18 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B+4) | 8 weeks, 6 months
  Designed to assess health related quality of life in breast cancer. Consists of 37 items and respondents are asked to indicate on a scale from 0 (not at all) through 4 (very much). Composed by five factors: physical quality of life; social / family and social quality of life; emotional quality of life; functional quality of life; and other concerns. FACT-B+4 has shown to have good. (Brady et al., 1997; Belmonte Martinez et al., 2011)

SECONDARY OUTCOMES:
Change Brief Symptom Inventory [BSI-18] | 8 weeks, 6 months
  BSI-18 measures general psychological distress, which consists of 18 descriptions of physical and emotional complaints; respondents are asked to indicate on a scale from 0 (not at all) through 4 (very much) to what extent they are troubled by the complaints. This scale is composed by 3 factors: Somatization, which refers to the discomfort caused by the perception of physical symptoms and body dysfunction.BSI-18 has shown to have good psychometric properties (Derogatis, 2001; Andreu et al., 2008)
Change Self-Compassion Scale-Short Form (SCS-SF) | 8 weeks, 6 months
  Designed to assess common humanity, mindfulness, self-judgment, over-identification, isolation, self-kindness and overall self-compassion. Composed by 12 items in its short verssion rated on a Likert scale from 1 (almost never) to 5 (almost always) with the total score derived by adding the means of each subscale together..SCS-SF has shown to have good (Raes, Pommier, Neff, & Van Gucht, 2011; Garcia-Campayo et al., 2014)
Change in The Compassion Scale (CS) | 8 weeks, 6 months
  A 24-item scale designed to assess compassion based on the six factor model of Neff's Self-Compassion Scale (Neff, 2003). In this study only the Total Compassion Score was utilized.CS has shown to have good (Pommier, 2010)
Change in Five Facets of Mindfulness Questionnaire - short form (FFMQ-SF) | 8 weeks, 6 months
  Measures participant's Mindfuless states and traits in daily life. It consists of 20 items rated on a scale ranging from 1 (never or very rarely true) to 5 (very often or always true). Itassess five factors of mindfulness: Observe, Describe,Acting with awareness, Non-judging of inner experience,and Non-reactivity to inner experience. FFMQ has shown to have good ((Tran, Glück, & Nader, 2013; Tran et al., 2014).
Change in Fear of Cancer Recurrence Inventory (FCRI) | 8 weeks to six months
  Designed to assess psychological stress and functional difficulties linked to cancer recurrence fear. Consists of 42-items that constitue seven components. In this study we only used 4 factors:(1) Triggers; (2) Psychological Distress; (3) Coping strategies; and (4) Insight. FCRI has shown to have good (Simard & Savard, 2009).

OTHER OUTCOMES:
High attendance (6 sessions) with protocol (CBCT® Evaluation Survey) | 8 weeks
  Designed to assess acceptance and adherence to the CBCT® Program. It consists of 20 items that evaluate: (1) attendance, (2) time (minutes) of home practice, (3) whether participants practiced with audio recordings or not, (4) frequency of practice, (5) whether participants intend to attend to future CBCT® Program courses or not,(6)& whether participants would recommend CBCT® Program or not, (7) satisfaction with CBCT® Program instructor's performance and (8) whether participants intend to continue with daily practice at home.
High minutes of home practice (CBCT® Evaluation Survey) | 8 weeks
  Designed to assess acceptance and adherence to the CBCT® Program. It consists of 20 items that evaluate: (1) attendance, (2) time (minutes) of home practice, (3) whether participants practiced with audio recordings or not, (4) frequency of practice, (5) whether participants intend to attend to future CBCT® Program courses or not,(6)& whether participants would recommend CBCT® Program or not, (7) satisfaction with CBCT® Program instructor's performance and (8) whether participants intend to continue with daily practice at home.
High percentage of home practice with recordings (CBCT® Evaluation Survey) | 8 weeks
  Designed to assess acceptance and adherence to the CBCT® Program. It consists of 20 items that evaluate: (1) attendance, (2) time (minutes) of home practice, (3) whether participants practiced with audio recordings or not, (4) frequency of practice, (5) whether participants intend to attend to future CBCT® Program courses or not,(6)& whether participants would recommend CBCT® Program or not, (7) satisfaction with CBCT® Program instructor's performance and (8) whether participants intend to continue with daily practice at home.
High frequency of practice between sessions (CBCT® Evaluation Survey) | 8 weeks
  Designed to assess acceptance and adherence to the CBCT® Program. It consists of 20 items that evaluate: (1) attendance, (2) time (minutes) of home practice, (3) whether participants practiced with audio recordings or not, (4) frequency of practice, (5) whether participants intend to attend to future CBCT® Program courses or not,(6) whether participants would recommend CBCT® Program or not, (7) satisfaction with CBCT® Program instructor's performance and (8) whether participants intend to continue with daily practice at home.
High percentage of intention to attend to future CBCT® Program courses (CBCT® Evaluation Survey) | 8 weeks
  Designed to assess acceptance and adherence to the CBCT® Program. It consists of 20 items that evaluate: (1) attendance, (2) time (minutes) of home practice, (3) whether participants practiced with audio recordings or not, (4) frequency of practice, (5) whether participants intend to attend to future CBCT® Program courses or not,(6)whether participants would recommend CBCT® Program or not, (7) satisfaction with CBCT® Program instructor's performance and (8) whether participants intend to continue with daily practice at home.
High recommendation rate of CBCT® Program courses (CBCT® Evaluation Survey) | 8 weeks
  Designed to assess acceptance and adherence to the CBCT® Program. It consists of 20 items that evaluate: (1) attendance, (2) time (minutes) of home practice, (3) whether participants practiced with audio recordings or not, (4) frequency of practice, (5) whether participants intend to attend to future CBCT® Program courses or not,(6)whether participants would recommend CBCT® Program or not, (7) satisfaction with CBCT® Program instructor's performance and (8) whether participants intend to continue with daily practice at home.
High satisfaction rate with CBCT® Program instructor's performance (CBCT® Evaluation Survey) | 8 weeks
  Designed to assess acceptance and adherence to the CBCT® Program. It consists of 20 items that evaluate: (1) attendance, (2) time (minutes) of home practice, (3) whether participants practiced with audio recordings or not, (4) frequency of practice, (5) whether participants intend to attend to future CBCT® Program courses or not,(6)whether participants would recommend CBCT® Program or not, (7) satisfaction with CBCT® Program instructor's performance and (8) whether participants intend to continue with daily practice at home.
High intention rate to continue with daily practice at home (CBCT® Evaluation Survey) | 8 weeks
  Designed to assess acceptance and adherence to the CBCT® Program. It consists of 20 items that evaluate: (1) attendance, (2) time (minutes) of home practice, (3) whether participants practiced with audio recordings or not, (4) frequency of practice, (5) whether participants intend to attend to future CBCT® Program courses or not,(6)whether participants would recommend CBCT® Program or not, (7) satisfaction with CBCT® Program instructor's performance and (8) whether participants intend to continue with daily practice at home.

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Gonzalez-Hernandez, Principal Investigator — Universitat de València; Rebeca Diego Pedro, PhD, Principal Investigator — Universitat de València; Rocío Romero Retes, PhD, Principal Investigator — Fundación Instituto Valenciano de Oncología; Daniel Campos Bacas, PhD, Principal Investigator — Universitat Jaume I; Lobsang Tenzin Negi aka Satya Dev Negi, PhD, Principal Investigator — Emory University / Emory-Tibet Partnership; Diana Burichka, Principal Investigator — Universitat de València
Locations (1):
- Fundación Instituto Valenciano de Oncología, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Rosenfeld, B., Krivo, S., Breitbart, W., & Chochinov, H. M. (2000). Suicide, assisted suicide, and euthanasia in the terminally ill.
- [Background] Rosedale M. Survivor loneliness of women following breast cancer. Oncol Nurs Forum. 2009 Mar;36(2):175-83. doi: 10.1188/09.ONF.175-183. PMID 19273406
- [Background] Pace TW, Negi LT, Dodson-Lavelle B, Ozawa-de Silva B, Reddy SD, Cole SP, Danese A, Craighead LW, Raison CL. Engagement with Cognitively-Based Compassion Training is associated with reduced salivary C-reactive protein from before to after training in foster care program adolescents. Psychoneuroendocrinology. 2013 Feb;38(2):294-9. doi: 10.1016/j.psyneuen.2012.05.019. Epub 2012 Jul 3. PMID 22762896
- [Background] Pace TW, Negi LT, Adame DD, Cole SP, Sivilli TI, Brown TD, Issa MJ, Raison CL. Effect of compassion meditation on neuroendocrine, innate immune and behavioral responses to psychosocial stress. Psychoneuroendocrinology. 2009 Jan;34(1):87-98. doi: 10.1016/j.psyneuen.2008.08.011. Epub 2008 Oct 4. PMID 18835662
- [Background] Negi, L. T. (2103). Emory compassion meditation protocol: Cognitively-based compassion training manualemory compassion meditation protocol: Cognitively-based compassion training manual. Atlanta: Emory University.
- [Background] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Background] Moorey, S., Greer, S., & Greer, S. (2002). Cognitive behaviour therapy for people with cancer Oxford University Press Oxford.
- [Background] Moorey, S. (2007). Breast cancer and body image. The Female Body in Mind: The Interface between the Female Body and Mental Health, , 72.
- [Background] Matthews H, Grunfeld EA, Turner A. The efficacy of interventions to improve psychosocial outcomes following surgical treatment for breast cancer: a systematic review and meta-analysis. Psychooncology. 2017 May;26(5):593-607. doi: 10.1002/pon.4199. Epub 2016 Aug 2. PMID 27333194
- [Background] Kok BE, Coffey KA, Cohn MA, Catalino LI, Vacharkulksemsuk T, Algoe SB, Brantley M, Fredrickson BL. How positive emotions build physical health: perceived positive social connections account for the upward spiral between positive emotions and vagal tone. Psychol Sci. 2013 Jul 1;24(7):1123-32. doi: 10.1177/0956797612470827. Epub 2013 May 6. PMID 23649562
- [Background] Jennings, P. A., Foltz, C., Snowberg, K. E., Sim, H., & Kemeny, M. E. (2011). The influence of mindfulness and emotion skills training on teachers' classrooms: The effects of the cultivating emotional balance training. Online Submission,
- [Background] Hofmann SG, Grossman P, Hinton DE. Loving-kindness and compassion meditation: potential for psychological interventions. Clin Psychol Rev. 2011 Nov;31(7):1126-32. doi: 10.1016/j.cpr.2011.07.003. Epub 2011 Jul 26. PMID 21840289
- [Background] Gilbert, P. (2010). An introduction to the theory & practice of compassion focused therapy and compassionate mind training for shame based difficulties. Retrieved
- [Background] García-Campayo, J., Navarro-Gil, M., & Demarzo, M. (2016). Attachment-based compassion therapy. Mindfulness & Compassion,
- [Background] Garcia-Campayo J, Demarzo M, Shonin E, Van Gordon W. How Do Cultural Factors Influence the Teaching and Practice of Mindfulness and Compassion in Latin Countries? Front Psychol. 2017 Jul 11;8:1161. doi: 10.3389/fpsyg.2017.01161. eCollection 2017. No abstract available. PMID 28744247
- [Background] García-Campayo, J., Cebolla, A., & Demarzo, M. (2016). La ciencia de la compasión (1ª ed.). Madrid: Alianza.
- [Background] Galceran J, Ameijide A, Carulla M, Mateos A, Quiros JR, Rojas D, Aleman A, Torrella A, Chico M, Vicente M, Diaz JM, Larranaga N, Marcos-Gragera R, Sanchez MJ, Perucha J, Franch P, Navarro C, Ardanaz E, Bigorra J, Rodrigo P, Bonet RP; REDECAN Working Group. Cancer incidence in Spain, 2015. Clin Transl Oncol. 2017 Jul;19(7):799-825. doi: 10.1007/s12094-016-1607-9. Epub 2017 Jan 16. PMID 28093701
- [Background] Fredrickson BL, Cohn MA, Coffey KA, Pek J, Finkel SM. Open hearts build lives: positive emotions, induced through loving-kindness meditation, build consequential personal resources. J Pers Soc Psychol. 2008 Nov;95(5):1045-1062. doi: 10.1037/a0013262. PMID 18954193
- [Background] Dodds SE, Pace TW, Bell ML, Fiero M, Negi LT, Raison CL, Weihs KL. Feasibility of Cognitively-Based Compassion Training (CBCT) for breast cancer survivors: a randomized, wait list controlled pilot study. Support Care Cancer. 2015 Dec;23(12):3599-608. doi: 10.1007/s00520-015-2888-1. Epub 2015 Aug 16. PMID 26275769
- [Background] Demarzo MM, Cebolla A, Garcia-Campayo J. The implementation of mindfulness in healthcare systems: a theoretical analysis. Gen Hosp Psychiatry. 2015 Mar-Apr;37(2):166-71. doi: 10.1016/j.genhosppsych.2014.11.013. Epub 2014 Dec 10. PMID 25660344
- [Background] Cebolla A, Campos D, Galiana L, Oliver A, Tomas JM, Feliu-Soler A, Soler J, Garcia-Campayo J, Demarzo M, Banos RM. Exploring relations among mindfulness facets and various meditation practices: Do they work in different ways? Conscious Cogn. 2017 Mar;49:172-180. doi: 10.1016/j.concog.2017.01.012. Epub 2017 Feb 20. PMID 28214767
- [Background] Carson JW, Keefe FJ, Lynch TR, Carson KM, Goli V, Fras AM, Thorp SR. Loving-kindness meditation for chronic low back pain: results from a pilot trial. J Holist Nurs. 2005 Sep;23(3):287-304. doi: 10.1177/0898010105277651. PMID 16049118
- [Background] Carlson LE, Speca M, Faris P, Patel KD. One year pre-post intervention follow-up of psychological, immune, endocrine and blood pressure outcomes of mindfulness-based stress reduction (MBSR) in breast and prostate cancer outpatients. Brain Behav Immun. 2007 Nov;21(8):1038-49. doi: 10.1016/j.bbi.2007.04.002. Epub 2007 May 22. PMID 17521871
- [Background] Burgess C, Cornelius V, Love S, Graham J, Richards M, Ramirez A. Depression and anxiety in women with early breast cancer: five year observational cohort study. BMJ. 2005 Mar 26;330(7493):702. doi: 10.1136/bmj.38343.670868.D3. Epub 2005 Feb 4. PMID 15695497
- [Background] Buick, D. L., Petrie, K. J., Booth, R., Probert, J., Benjamin, C., & Harvey, V. (2000). Emotional and functional impact of radiotherapy and chemotherapy on patients with primary breast cancer. Journal of Psychosocial Oncology, 18(1), 39-62.
- [Background] Bower JE, Ganz PA, Desmond KA, Rowland JH, Meyerowitz BE, Belin TR. Fatigue in breast cancer survivors: occurrence, correlates, and impact on quality of life. J Clin Oncol. 2000 Feb;18(4):743-53. doi: 10.1200/JCO.2000.18.4.743. PMID 10673515
- [Background] Bleiker EM, Pouwer F, van der Ploeg HM, Leer JW, Ader HJ. Psychological distress two years after diagnosis of breast cancer: frequency and prediction. Patient Educ Couns. 2000 Jun;40(3):209-17. doi: 10.1016/s0738-3991(99)00085-3. PMID 10838000
- [Background] Bellver, A., Sánchez-Cánovas, J., Santaballa, A., Munárriz, B., Pérez-Fidalgo, J. A., & Montalar, J. (2009). Mujeres con cáncer de mama: Evaluación del afecto positivo y negativo y valoración de un programa de intervención psicológica en el ámbito hospitalario. Psicooncología, 6(1), 139.
- [Background] Bartley, T. (2011). Mindfulness-based cognitive therapy for cancer John Wiley & Sons.
- [Background] Baer, R. A., Lykins, E. L., & Peters, J. R. (2012). Mindfulness and self-compassion as predictors of psychological wellbeing in long-term meditators and matched nonmeditators. The Journal of Positive Psychology, 7(3), 230-238.
- [Background] Andersen BL, Farrar WB, Golden-Kreutz DM, Glaser R, Emery CF, Crespin TR, Shapiro CL, Carson WE 3rd. Psychological, behavioral, and immune changes after a psychological intervention: a clinical trial. J Clin Oncol. 2004 Sep 1;22(17):3570-80. doi: 10.1200/JCO.2004.06.030. PMID 15337807
- [Result] Zabora J, BrintzenhofeSzoc K, Curbow B, Hooker C, Piantadosi S. The prevalence of psychological distress by cancer site. Psychooncology. 2001 Jan-Feb;10(1):19-28. doi: 10.1002/1099-1611(200101/02)10:13.0.co;2-6. PMID 11180574
- [Result] Thewes B, Butow P, Bell ML, Beith J, Stuart-Harris R, Grossi M, Capp A, Dalley D; FCR Study Advisory Committee. Fear of cancer recurrence in young women with a history of early-stage breast cancer: a cross-sectional study of prevalence and association with health behaviours. Support Care Cancer. 2012 Nov;20(11):2651-9. doi: 10.1007/s00520-011-1371-x. Epub 2012 Feb 11. PMID 22328003
- [Result] Thewes B, Brebach R, Dzidowska M, Rhodes P, Sharpe L, Butow P. Current approaches to managing fear of cancer recurrence; a descriptive survey of psychosocial and clinical health professionals. Psychooncology. 2014 Apr;23(4):390-6. doi: 10.1002/pon.3423. Epub 2013 Nov 1. PMID 24307136
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Result] Sansó, N., Galiana, L., Cebolla, A., Oliver, A., Benito, E., & Ekman, E. (2017). Cultivating emotional balance in professional caregivers: A pilot intervention. Mindfulness, , 1-9.
- [Derived] Gonzalez-Hernandez E, Romero R, Campos D, Burychka D, Diego-Pedro R, Banos R, Negi LT, Cebolla A. Cognitively-Based Compassion Training (CBCT(R)) in Breast Cancer Survivors: A Randomized Clinical Trial Study. Integr Cancer Ther. 2018 Sep;17(3):684-696. doi: 10.1177/1534735418772095. Epub 2018 Apr 22. PMID 29681185
- See also: Weiss, M. C. (2017). U.S. breast cancer statistics. — http://www.breastcancer.org/symptoms/understand_bc/statistics